CLINICAL TRIAL: NCT04433923
Title: Aluminium Foil as an Adjuvant to Phototherapy for Pathological Unconjugated Hyperbilirubinaemia in Full Term Infants: Randomised Control Trial
Brief Title: Aluminium Foil as an Adjuvant to Phototherapy for Pathological Unconjugated Hyperbilirubinaemia in Full Term Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Abd Elazeez Attala Shabaan, Professor, Mansoura University
Purpose: Treatment
Other Study IDs: MansouraU004
Record Dates: First submitted 2020-06-13; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Neonatal Jaundice
MeSH Terms: conditions — Jaundice, Neonatal | interventions — Phototherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No

ARMS (2):
- GROUP1 (Active Comparator): Phototherapy with aluminum foil
  Interventions: Device: Phototherapy with aluminum foil
- GROUP2 (Placebo Comparator): Phototherapy without aluminum foil
  Interventions: Device: Phototherapy without aluminum foil

INTERVENTIONS:
Device: Phototherapy with aluminum foil
  Arms: GROUP1
Device: Phototherapy without aluminum foil
  Arms: GROUP2

SUMMARY:
prospective single center pilot randomized open label clinical trial, conducted at the Neonatal care unit of Mansoura University Children's To assess the efficacy and safety of aluminum foil use in combination with phototherapy compared with phototherapy alone for pathological unconjugated hyperbilirubinaemia in full term newborn We enrolled 234 infants in the study who fulfilled the inclusion criteria and were randomly assigned to treatment groups, either conventional phototherapy with aluminum foil or conventional phototherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Appropriate for gestational age full-term infants with pathological unconjugated hyperbilirubinaemia who are candidate for photo therapy according to American academy guidelines

Exclusion Criteria:

* Preterm infants, newborn infant with congenital malformations, conjugated hyperbilirubinamia, small for gestational age, in need of exchange transfusion, and skin abrasions or infections

Max Age: 28 Days | Sex: All
Age Groups: Child
Dates: Start 2016-06-01; Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Total serum bilirubin | 8 hours of treatment
  measurement of Total serum bilirubin (mg/dl)
Total serum bilirubin | 24 hours of treatment
  measurement of Total serum bilirubin (mg/dl)
Total serum bilirubin | 48 hours of treatment
  measurement of Total serum bilirubin (mg/dl)

SECONDARY OUTCOMES:
duration of photo therapy | average 48 hours
  duration of photo therapy in hours

IPD SHARING:
Plan to Share IPD: Undecided